CLINICAL TRIAL: NCT04264559
Title: The Heat Transport Characteristics of the Heart and Lung Meridians: A Study of CSAP Patients and Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019ZY009-MERIDIAN
Record Dates: First submitted 2020-02-08; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Chronic Stable Angina Pectoris
Keywords: stable angina pectoris; meridian; infrared thermal imaging
MeSH Terms: conditions — Angina, Stable | interventions — Moxibustion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy control group (Other): This group will include 40 healthy adults.
  Interventions: Diagnostic Test: Infrared thermal imaging
- CSAP group (Other): This study will include 40 patients with chronic stable angina pectoris (CSAP).
  Interventions: Diagnostic Test: Infrared thermal imaging
- Healthy intervention group (Experimental): This group will include 40 healthy adults. They will receive moxibustion intervention.
  Interventions: Diagnostic Test: Infrared thermal imaging; Procedure: Moxibustion

INTERVENTIONS:
Diagnostic Test: Infrared thermal imaging — A thermal imager is used to record thermal images.The baseline temperature of relevant acupoints or sites on the Heart and Lung meridians will be measured.
Procedure: Moxibustion — Two sessions of moxibustion intervention will be performed in the Heart meridian and Lung meridian successively. During moxibustion, the temperature change of relevant acupoints or sites in the Heart and Lung meridians will be measured by infrared thermal imaging.
  * Intervention in the Heart meridian: moxibustion will be performed in acupoint HT3 of the Heart meridian for 15 minutes.
  * Intervention in the Lung meridian: moxibustion will be performed in acupoint LU5 of the Lung meridian for 15 minutes.
  Arms: Healthy intervention group

SUMMARY:
Although some important progresses were made in the field of the meridian research, no breakthroughs have been achieved. Besides,there are some problems in meridian researches. Particularly, previous research of meridian phenomena involved lots of subjective elements and outcomes.Researches that use modern scientific techniques to investigate the biological characteristics of meridian phenomenon are urgently needed. Therefore, this study is designed to assess the heat transport characteristics of the Heart and Lung meridians by infrared thermal imaging (ITI). Thus, the biological characteristics of meridian phenomena could be presented objectively in a scientific methodology

DETAILED DESCRIPTION:
This study will include 40 patients with chronic stable angina pectoris (CSAP), and 80 healthy adults. Infrared thermal imaging (ITI) examination will be adopted to assess the heat transport characteristics of the Heart and Lung meridians and investigate the specificity for the meridian-visceral correlation and site-to-site correlation between two specific meridians.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for CSAP patients

* Patients should meet the diagnostic criteria of coronary heart disease, which includes the following items: 1)confirmed old myocardial infarction (MI), or a history of percutaneous coronary intervention(PCI), or coronary artery bypass grafting; 2)50% or more luminal stenosis in at least one coronary artery or major branch segment confirmed by coronary angiogram or CT angiography; 3) myocardial ischemia indicted by exercise stress radionuclide myocardial imaging; 4) treadmill exercise testing is positive (for male patients);
* Patients should meet the diagnostic criteria of CSAP and the Canadian Cardiovascular Society(CCS) classification for CSAP is level II or III;
* The medical history of CSAP is more than 3 months with attacks occurring at least twice weekly in the last month;
* 35≤age ≤75 years, male or female;
* Patients have clear consciousness and could communicate with others normally;
* Patients could understand the full study protocol and written informed consent is signed.

Inclusion criteria for healthy adults

* Healthy volunteers who could provide a recent medical examination report to confirm they have not any cardiovascular and respiratory disease;
* age≥20 years, male or female;
* Participants have clear consciousness and could communicate with others normally;
* Participants could understand the full study protocol and written consent is signed.

Exclusion Criteria:

Exclusion criteria for CSAP patients

* Patients have acute coronary syndrome and severe arrhythmias;
* Patients' chest pain is caused by valvular heart disease, hypertrophic cardiomyopathy and dilated cardiomyopathy;
* Patients' chest pain is caused by non-cardiac disease;
* Patients have concomitant lung diseases;
* Patients have serious concomitant conditions and fail to treat them effectively, such as diseases of the digestive, urinary, respiratory, hematological and nervous system;
* Patients have mental illness, severe depression, alcohol dependence or history of drug abuse;
* Pregnant or lactating patients;
* Patients are participating in other trials.

Exclusion criteria for healthy adults

* Participants have mental illness, severe depression, alcohol dependence or history of drug abuse;
* Pregnant or lactating participants ;
* Participants are participating in other trials.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Temperature change of relevant acupoints or sites | Baseline, 15 minutes during moxibustion, 5 minutes after stopping moxibustion.
  Infrared thermal imaging examination is used to assess temperature change of relevant acupoints or sites of the Heart and Lung meridians

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China